CLINICAL TRIAL: NCT04738591
Title: Feasibility Study Through a Phase II Randomized Clinical Trial of an Intervention Based on Short Message System (SMS) to Promote Adherence to Antidiabetic Medication and Healthy Lifestyles in Patients With Type 2 Diabetes Mellitus
Brief Title: mHealth Intervention to Support Diabetes Medication Adherence (Pilot Study)
Acronym: DIABE-TEXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RTI2018-096935-A-I00_pilot; IB 43/20/20 PI (Other: Research Ethics Committee of the Balearic Islands)
Record Dates: First submitted 2021-01-28; First posted 2021-02-04 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Medication; Adherence; Glycaemic control; Healthy lifestyle; mHealth; SMS
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIABE-TEXT (Experimental): Participants allocated to the intervention group will receive text messages in their mobile phones with content about diabetes management, general information about diabetes, medicines, diet and physical activity recommendations and motivational prompts to engage participants in a healthy lifestyle and a good adherence to medication plan. They will also receive reminders for healthcare visits, drug dispensation from the pharmacy and updated results from blood test records.
  Interventions: Device: DIABE-TEXT
- Usual care (No Intervention): Participants allocated to the control group will not receive any intervention apart from usual care.

INTERVENTIONS:
Device: DIABE-TEXT — Participants will receive daily (from monday to friday) text messages in their mobile phones during three months.
  Arms: DIABE-TEXT

SUMMARY:
This study aims at evaluating the feasibility of an intervention based on the use of a mobile-device based system delivering automated, tailored brief text messages to offer support for medicine use and lifestyle recommendations alongside usual care to people with type 2 diabetes.

DETAILED DESCRIPTION:
A list of patients registered in primary care centers of the Balearic Islands and potentially meeting the eligibility criteria will be obtained from electronic health records (EHRs). A research assistant will contact the potential participants via phone to invite them to the study and confirm eligibility. All eligible participants will complete informed consent followed by baseline assessment over the phone before randomization. Participants will be randomly allocated using a computer-generated randomization sequence. All participants will continue with their usual diabetes care including all medical visits, tests, and diabetes support programs throughout the study. In addition, the intervention group will receive the text messaging intervention. Control participants will receive usual care only. After three months of follow-up, all participants will complete post-intervention assessments via phone interview. Data on glycemic control (HbA1c) at baseline and post-intervention will be extracted from EHRs, as according to the protocol used for primary care providers in the Balearic Islands, patients with poor glycemic control (HbA1c >8% ) must request an HbA1c determination every six months. Results of the most recent determination will be extracted from electronic medical records. For those patients with no recorded HbA1c within the previous three months, the research assistant will contact the primary care center and the patient to arrange blood test analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients registered in the Public Health Service of the Balearic Islands
* With type 2 diabetes
* At least one prescription of an oral glucose-lowering drug
* With results of HbA1C>8% from 3 months prior to recruitment.

Exclusion Criteria:

* Younger than 18 years old
* With insulin treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ignacio Ricci-Cabello, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Background] Arambepola C, Ricci-Cabello I, Manikavasagam P, Roberts N, French DP, Farmer A. The Impact of Automated Brief Messages Promoting Lifestyle Changes Delivered Via Mobile Devices to People with Type 2 Diabetes: A Systematic Literature Review and Meta-Analysis of Controlled Trials. J Med Internet Res. 2016 Apr 19;18(4):e86. doi: 10.2196/jmir.5425. PMID 27095386
- [Background] Farmer AJ, McSharry J, Rowbotham S, McGowan L, Ricci-Cabello I, French DP. Effects of interventions promoting monitoring of medication use and brief messaging on medication adherence for people with Type 2 diabetes: a systematic review of randomized trials. Diabet Med. 2016 May;33(5):565-79. doi: 10.1111/dme.12987. Epub 2015 Nov 17. PMID 26470750
- [Derived] Zamanillo-Campos R, Fiol-deRoque MA, Serrano-Ripoll MJ, Mira-Martinez S, Ricci-Cabello I. Development and evaluation of DiabeText, a personalized mHealth intervention to support medication adherence and lifestyle change behaviour in patients with type 2 diabetes in Spain: A mixed-methods phase II pragmatic randomized controlled clinical trial. Int J Med Inform. 2023 Aug;176:105103. doi: 10.1016/j.ijmedinf.2023.105103. Epub 2023 May 22. PMID 37267809

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DIABE-TEXT | Usual Care
Started | 96 | 111
Completed | 89 | 90
Not Completed | 7 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DIABE-TEXT | Usual Care | Total
Number analyzed (Participants) | 96 | 111 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10) | 61 (12) | 62 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 61 | 74 | 135
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
HbA1c (%), Continuous [Mean (Standard Deviation); unit: Percentage of HbA1c] | 9 (1) | 9.1 (1.3) | 9 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Glycated Hemoglobin (HbA1C)
Description: HbA1c was extracted as percentage which is calculated following the standard formulae [HbA1c(%)=(HbA1c(mmol/mol)+23.5)/10.93] based on its concentration in blood samples. It identifies average plasma glucose concentration.
Time Frame: Baseline and post-intervention at 3 months
Population: The number analyzed post-intervention differs from overall number analyzed because of losses to follow-up.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | DIABE-TEXT | Usual Care
Number analyzed (Participants) | 96 | 111
Percentage of HbA1c
  Baseline | 9 (1) | 9.1 (1.3)
  Post-intervention | 7.7 (1.3) | 7.6 (1.2)

2. Secondary Outcome: Number of Participants Classified as Adherent Based on Self-reporteAdherence to Antidiabetic Medication (7 Items ad Hoc Questionnaire)
Description: Number of participants classified as adherent based on Self-reported adherence to glucose medications was measured with a 7-items ad hoc questionnaire adapted from Chaves-Torres et al. for people with type 2 diabetes. Participants who obtained 7 points were considered adherent while the ones with < 7 points were non-adherent.
Time Frame: Baseline and post-intervention at 3 months
Population: The number analyzed post-intervention differs from overall number analyzed at baseline because of lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | DIABE-TEXT | Usual Care
Number analyzed (Participants) | 96 | 111
Participants
  Baseline | 72 | 76
  Post-intervention: number analyzed (Participants) | 89 | 90
  Post-intervention | 73 | 62

3. Secondary Outcome: Enrolment or Recruitment Rate
Description: (Patients enroled/ Total Eligible patients) x 100 percent
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: People meeting eligibility criteria for inclusion in the study
Arm/Group | Eligible Participants
Number analyzed (Participants) | 444
Participants | 207

4. Secondary Outcome: Retention Rate
Description: (Patients who finish follow-up/Total recruited) x 100 percent
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | DIABE-TEXT | Usual Care
Number analyzed (Participants) | 96 | 111
Participants | 89 | 90

5. Other Pre Specified Outcome: 14-point Mediterranean Diet Adherence Screener (MEDAS-14)
Description: The 14-point Mediterranean Diet Adherence Screener (MEDAS-14) questionnaire was registered at baseline and post-intervention. Participants were classified as low adherents (≤5), moderate adherents (6 to 9 points) or high adherents (≥10 points) according to the results obtained that can range between 1 to 14 points. After that, we joined moderate adherents with high adherents and tagged them as adherents to the Mediterranean Diet, while low adherents were considered non-adherents to the Mediterranean diet. Therefore, we presented the number of participants adherent to the MediterraneanDiet. A higher score means a higher adherence to Mediterranean diet. Results obtained through the website from the Public Health System of the Balearic Islands: https://apps.caib.es/plasalutfront/formularios/dieta/dieta.xhtml
Time Frame: Baseline and post-intervention at 3 months
Population: The number analyzed post-intervention differs from overall number analyzed at baseline because of lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | DIABE-TEXT | Usual Care
Number analyzed (Participants) | 96 | 111
Participants
  Baseline | 49 | 55
  Post-intervention: number analyzed (Participants) | 89 | 90
  Post-intervention | 53 | 43

6. Other Pre Specified Outcome: Being Adherent to Physical Activity Recommendations Based on Having Moderate or High Levels of Physical Activity Resulted From the International Physical Activity Questionnaire (IPAQ)
Description: A 6-items adapted from the short version of the International Physical Activity Questionnaire (IPAQ) (11) was registered at baseline and post-intervention. Participants were classified as having a low, moderate or high level of physical activity based on metabolic equivalent of task (METs) calculation. After that, we joined the participants that presented moderate or high level of physical activity and tagged them as adherents to Physical Activity recommendations, while having low levels of Physical Activity was considered as being non-adherent to the Physical Activity Recommendations. Therefore, we presented the number of participants adherent to the Physical Activity Recommendations.
  We used the available tool from the Public Health System of the Balearic Islands: https://apps.caib.es/plasalutfront/formularios/ipaq/ipaq.xhtml
Time Frame: Baseline and post-intervention at 3 months
Population: The number analyzed post-intervention differs from overall number analyzed at baseline because of lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | DIABE-TEXT | Usual Care
Number analyzed (Participants) | 96 | 111
Participants
  Baseline | 56 | 55
  Post-intervention: number analyzed (Participants) | 89 | 90
  Post-intervention | 62 | 52

ADVERSE EVENTS:
Time Frame: 3 months
Description: All-cause mortality and serious adverse events were not assessed; therefore, the number of affected participants cannot be reported accurately.
Arm/Group | DIABE-TEXT | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/96 | 0/111
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DIABE-TEXT (N=96) | Usual Care (N=111)
Feeling emotionally distressed (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
First, rather than ordering laboratory tests to measure HbA1c, we extracted this data from electronic clinical records. Second, we used an ad hoc questionnaire to measure medication adherence. Finally, although 99% of the SMS messages were successfully delivered, and 96% of the participants stated that they received and read the messages as intended, we were not able to track the number of messages actually opened by the participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT04738591/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT04738591/ICF_001.pdf